CLINICAL TRIAL: NCT03898167
Title: A Randomized Controlled Trial of Mailed Self-Sample HPV Testing to Increase Cervical Cancer Screening Participation Among Minority/Underserved Women in an Integrated Safety Net Healthcare System
Brief Title: Prospective Evaluation of Self-Testing to Increase Screening
Acronym: PRESTIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Jane Montealegre, Associate Professor, M.D. Anderson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: H-44944; R01MD013715 (NIH); R01MD013715-04S2 (NIH)
Record Dates: First submitted 2019-03-29; First posted 2019-04-01 (Actual); Results first posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Cervical Cancer; Human Papillomavirus Infection
Keywords: Screening; Human Papillomavirus Infection; Self-Testing
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections | interventions — Patient Navigation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Telephone Recall (Active Comparator): Participants receive a scripted telephone recall from a trained patient navigator on behalf of Harris Health System.
  Interventions: Behavioral: Telephone Recall
- Mailed HPV Self-Sampling Kit (Experimental): Participants receive a scripted telephone recall from a patient navigator on behalf of Harris Health System and receive a mailed HPV self-sampling kit with a pre-paid return envelope.
  Interventions: Behavioral: Telephone Recall; Behavioral: Mailed HPV Self-Sampling Kit
- Mailed HPV Self-Sampling Kit + Patient Navigation (Experimental): Participants receive a scripted telephone recall and mailed self-sampling kit with a pre-paid return envelope. Within 3-5 days of the kit's mail-out, participants will receive a telephone call from a patient navigator to provide one-on-one education.
  Interventions: Behavioral: Telephone Recall; Behavioral: Mailed HPV Self-Sampling Kit; Behavioral: Patient Navigation

INTERVENTIONS:
Behavioral: Telephone Recall — Participants receive a scripted telephone recall from a trained patient navigator.
Behavioral: Mailed HPV Self-Sampling Kit — Participants receive a mailed kit that allows them to self-collect a cervical sample in their home and return it to a laboratory for human papillomavirus (HPV) testing.
  Arms: Mailed HPV Self-Sampling Kit; Mailed HPV Self-Sampling Kit + Patient Navigation
Behavioral: Patient Navigation — Participant receives telephone call from patient navigator within 3-5 days of receipt of self-collection kit. Patient navigator provides one-on-one education on cervical cancer screening and self-collection of cervical sample.
  Arms: Mailed HPV Self-Sampling Kit + Patient Navigation

SUMMARY:
Regularly attending for Pap test cervical cancer screening in a clinic is often unfeasible and/or unacceptable to many women. This study evaluates if mailing and testing self-sampled kits for high-risk human papillomavirus (HPV) can cost-effectively increase screening participation among underserved minority women in a safety-net health system.

DETAILED DESCRIPTION:
Regularly attending for Pap test cervical cancer screening in a clinic is often unfeasible and/or unacceptable to many women. Using mailed self-sampling kits to test for high-risk human papillomavirus (HPV), the virus that causes cervical cancer, may overcome multiple barriers to clinic-based screening. This study is a randomized controlled trial to compare the effectiveness of three outreach interventions to increase primary screening participation and clinical follow-up among underscreened women a in a safety net health system. The three strategies that will be evaluated are: 1) telephone recall; 2) telephone recall with mailed self-sample HPV testing kits; and 3) telephone recall with mailed self-sample HPV testing kits and patient navigation.

ELIGIBILITY:
Inclusion Criteria:

* no history of hysterectomy or cervical cancer
* no Pap test in the past 3.5 years or Pap/HPV co-test in the past 5.5 years
* patient of Harris Health System in Harris County (Houston), Texas
* have at least 2 visits to ambulatory care within Harris Health System in the past 5 years
* be currently enrolled in a healthcare coverage or financial assistance plan accepted by Harris Health System or have been enrolled in a Harris Health coverage plan in the past 12 months

Exclusion Criteria:

* no valid telephone contact information
* unable to communicate in English or Spanish*
* currently pregnant
* history of cervical dysplasia in the past 3.5 years

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 2474 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2025-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane R Montealegre, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- Harris Health System, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared on primary and secondary outcomes. The PI will ensure all mechanisms used to share data will include proper plans and safeguards for the protection of privacy, confidentiality, and security for data dissemination and reuse (e.g., all data will be thoroughly de-identified and will not be traceable to a specific study participant).
Supporting Information: Study Protocol
Time Frame: De-identified data are available to study team members now and will be made available until primary, secondary and exploratory analyses are complete.
Access Criteria: Listed on IRB-approved protocol.

REFERENCES:
- [Background] Montealegre JR, Anderson ML, Hilsenbeck SG, Chiao EY, Cantor SB, Parker SL, Daheri M, Bulsara S, Escobar B, Deshmukh AA, Jibaja-Weiss ML, Zare M, Scheurer ME. Mailed self-sample HPV testing kits to improve cervical cancer screening in a safety net health system: protocol for a hybrid effectiveness-implementation randomized controlled trial. Trials. 2020 Oct 21;21(1):872. doi: 10.1186/s13063-020-04790-5. PMID 33087164
- [Background] Amboree TL, Parker SL, Bulsara S, Anderson ML, Schmeler KM, Chiao EY, Montealegre JR. Cervical cancer screening among English- and Spanish-speaking Hispanic women in an urban safety net health system, 2015-2020. BMC Womens Health. 2023 Jun 15;23(1):309. doi: 10.1186/s12905-023-02448-3. PMID 37316815
- [Result] Parker S, Deshmukh AA, Chen B, Lairson DR, Daheri M, Vernon SW, Montealegre JR. Perceived barriers to cervical cancer screening and motivators for at-home human papillomavirus self-sampling during the COVID-19 pandemic: Results from a telephone survey. Elife. 2023 May 26;12:e84664. doi: 10.7554/eLife.84664. PMID 37232493
- [Result] Parker SL, Amboree TL, Bulsara S, Daheri M, Anderson ML, Hilsenbeck SG, Jibaja-Weiss ML, Zare M, Schmeler KM, Deshmukh AA, Chiao EY, Scheurer ME, Montealegre JR. Self-Sampling for Human Papillomavirus Testing: Acceptability in a U.S. Safety Net Health System. Am J Prev Med. 2024 Mar;66(3):540-547. doi: 10.1016/j.amepre.2023.10.020. Epub 2023 Nov 5. PMID 37935320
- [Derived] Montealegre JR, Hilsenbeck SG, Bulsara S, Parker SL, Amboree TL, Anderson ML, Daheri M, Jibaja-Weiss ML, Schmeler KM, Deshmukh AA, Chiao EY, Scheurer ME. Self-Collection for Cervical Cancer Screening in a Safety-Net Setting: The PRESTIS Randomized Clinical Trial. JAMA Intern Med. 2025 Sep 1;185(9):1119-1127. doi: 10.1001/jamainternmed.2025.2971. PMID 40478588

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Trial enrollment began February 20,2020, then paused March 27, 2020, due to clinic closures and restrictions on human participant research following the declaration of the COVID-19 pandemic. Trial enrollment resumed August 3,2020 and continued through August 31, 2023.
Period: Overall Study
Arm/Group | Telephone Recall | Mailed HPV Self-Sampling Kit | Mailed HPV Self-Sampling Kit + Patient Navigation
Started | 828 | 828 | 818
Completed | 821 | 737 | 715
Not Completed | 7 | 91 | 103
Not completed — Terminated phone call early | 7 | 0 | 0
Not completed — Terminated phone call early or requested to not receive a kit | 0 | 91 | 103

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telephone Recall | Mailed HPV Self-Sampling Kit | Mailed HPV Self-Sampling Kit + Patient Navigation | Total
Number analyzed (Participants) | 828 | 828 | 818 | 2474
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 48 [39 to 57] | 49 [39 to 58] | 48 [39 to 57] | 49 [39 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 828 | 828 | 818 | 2474
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 578 | 548 | 529 | 1655
  Non-Hispanic Asian | 27 | 29 | 26 | 82
  Non-Hispanic Black or African American | 163 | 173 | 199 | 535
  Non-Hispanic White | 50 | 57 | 42 | 149
  Non-Hispanic Other or Unknown | 10 | 21 | 22 | 53
Region of Enrollment [Number; unit: participants]
  United States | 828 | 828 | 818 | 2474
Type of health care coverage [Count of Participants; unit: Participants]
  Private insurance | 246 | 246 | 245 | 737
  Publicly funded financial assistance plan | 476 | 461 | 451 | 1388
  Medicaid | 60 | 69 | 74 | 203
  Medicare | 27 | 30 | 23 | 80
  Other | 19 | 22 | 25 | 66

OUTCOME MEASURES:

1. Primary Outcome: Primary Screening Participation
Description: cervical cancer screening participation within 6 months, defined as return of a mailed HPV self-collection kit or attendance for clinic-based screening.
Time Frame: within 6 months of randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Telephone Recall | Mailed HPV Self-Sampling Kit | Mailed HPV Self-Sampling Kit + Patient Navigation
Number analyzed (Participants) | 828 | 828 | 818
Participants | 144 | 340 | 381
Statistical Analysis 1: Comparison: Telephone Recall vs Mailed HPV Self-Sampling Kit vs Mailed HPV Self-Sampling Kit + Patient Navigation; Bivariable tables, Pearson chi-square and Kruskal-Wallis nonparametric tests were used to compare demographic/health care characteristics by study group. Log binomial regression was used to calculate screening proportion, participation difference, and relative participation (calculated as relative risk), with 95% CIs. Overall participation difference and relative participation for SC and SC with patient navigation vs TR were calculated by combining numerators and denominators from each group; Test type: Other; 95% CIs were calculated; Relative Participation = 2.36, 95% CI 2-sided [1.99 to 2.80]

2. Secondary Outcome: Screening Tests Results
Description: Results of HPV test using self-collected samples (positive, negative, or inadequate)
Time Frame: within 6 months of randomization
Population: Participated in cervical cancer screening
Measure: Count of Participants; unit: Participants
Arm/Group | Telephone Recall | Mailed HPV Self-Sampling Kit | Mailed HPV Self-Sampling Kit + Patient Navigation
Number analyzed (Participants) | 144 | 340 | 381
Participants
  Positive | 6 | 38 | 49
  Negative | 138 | 288 | 312
  Inadequate | 0 | 14 | 20

3. Secondary Outcome: Completion of Clinical Follow-up Among Women With an Abnormal Screening Test Result
Description: Electronic medical record (EMR)-confirmed attendance for colposcopy among participants who had a positive test by clinic-based screening; EMR- confirmed attendance for colposcopy or subsequent clinic-based screening among those who had a positive test by self-sampling
Time Frame: Attendance to clinical follow up was assessed within 12 months of screening test result, up to 18 months post randomization.
Population: Participants with an abnormal screening result, including those received from a clinic-based screening or mailed HPV self-sampling kit.
Measure: Count of Participants; unit: Participants
Arm/Group | Telephone Recall | Mailed HPV Self-Sampling Kit | Mailed HPV Self-Sampling Kit + Patient Navigation
Number analyzed (Participants) | 6 | 36 | 48
Participants
  Attended follow up | 2 | 22 | 33
  Did not attend follow up | 4 | 14 | 15

ADVERSE EVENTS:
Time Frame: Within 6 months post randomization
Description: Study participants were asked to report any adverse events during the use of the HPV self-collection kit. Reported AEs were assessed within 6 months of randomization.**
  **AEs are for when participants are "on treatment" so would have been within 6 months post randomization.
Arm/Group | Telephone Recall | Mailed HPV Self-Sampling Kit | Mailed HPV Self-Sampling Kit + Patient Navigation
All-Cause Mortality (participants affected / at risk) | 0/828 | 0/828 | 0/818
Serious Adverse Events (participants affected / at risk) | 0/828 | 0/828 | 0/818
Other Adverse Events (participants affected / at risk) | 0/828 | 0/828 | 1/818
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telephone Recall (N=828) | Mailed HPV Self-Sampling Kit (N=828) | Mailed HPV Self-Sampling Kit + Patient Navigation (N=818)
Pain (General disorders) | 0 | 0 | 1 (1)

LIMITATIONS AND CAVEATS:
Participants knew self-collection was part of research study; trial overlapped with COVID-19 pandemic; patient navigators were unblinded; trial was not powered to test differences in follow-up; samples were tested using the non-FDA approved Aptima HPV test; FDA approved self-collection in clinical settings following completion of trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-25): https://cdn.clinicaltrials.gov/large-docs/67/NCT03898167/Prot_SAP_000.pdf